CLINICAL TRIAL: NCT00001039
Title: The Effect of Therapy on the Tissue Burden of Disseminated MAC Infection as Measured by Quantitative Bone Marrow Culture and Correlation With Quantitative Blood Culture in HIV-Infected Patients
Brief Title: Evaluation of Treatment for Mycobacterium Avium Complex (MAC) Infection in HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: DATRI 007; 11739 (Registry Identifier: DAIDS ES Registry ID)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Mycobacterium Avium-intracellulare Infection; HIV Infections
Keywords: Mycobacterium avium-intracellulare Infection; Drug Therapy, Combination; Ethambutol; Acquired Immunodeficiency Syndrome; Clarithromycin
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Ethambutol; Clarithromycin

INTERVENTIONS:
Drug: Ethambutol hydrochloride
Drug: Clarithromycin

SUMMARY:
To assess the feasibility of using culture and staining techniques to quantify tissue Mycobacterium avium Complex (MAC) burden in bone marrow. To correlate and compare changes in MAC bone marrow burden with quantitative MAC blood culture results at baseline and after 4 and 8 weeks of treatment.

MAC is easiest to detect in the blood, although doctors generally believe that MAC in blood is just "spill-over" from infection of other parts of the body. Traditionally, studies of potential treatments for MAC focus only on MAC changes in the blood. This study compares MAC changes in blood to those in bone marrow, which is another tissue where MAC is often found.

DETAILED DESCRIPTION:
MAC is easiest to detect in the blood, although doctors generally believe that MAC in blood is just "spill-over" from infection of other parts of the body. Traditionally, studies of potential treatments for MAC focus only on MAC changes in the blood. This study compares MAC changes in blood to those in bone marrow, which is another tissue where MAC is often found.

Patients receive both clarithromycin and ethambutol for 48 weeks; those who become intolerant to the study drugs may receive suggested substitute drugs (azithromycin and rifabutin). Patients receive a bone marrow biopsy at baseline and at either 4 or 8 weeks. Patients are evaluated at weeks 1, 2, 4, 6, 8, 12, 24, 36, and 48.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Any antiretroviral therapy that is approved or is available through an FDA-sanctioned treatment IND or treatment protocol.
* Primary or secondary PCP prophylaxis with TMP/SMX, dapsone, or aerosolized pentamidine, as well as approved therapies for other AIDS-related opportunistic infections not otherwise excluded.
* Erythromycin, interferon-alpha, and supportive care for any therapy-related toxicities as necessary.

Patients must have:

* HIV infection.
* Confirmed MAC bacteremia.
* Consent of parent or guardian if less than 18 years of age.

Exclusion Criteria

Concurrent Medication:

Excluded:

* MAC inhibitors, including aminoglycosides, quinolones, clofazimine, azithromycin (except when administered as a substitute drug), and rifamycins, during the first 24 weeks of the study.
* Immunomodulators (including colony-stimulating cytokines such as GM-CSF and G-CSF) other than those that are specifically allowed.
* Steroids in excess of physiologic replacement doses.
* Cytotoxic chemotherapy.

Patients with the following prior conditions are excluded:

* History of treatment-limiting intolerance or hypersensitivity to the study drugs or other macrolides.
* Changes on chest radiograph within 7 days prior to study entry, that are consistent with acute Pneumocystis carinii pneumonia, pulmonary tuberculosis, or other acute respiratory infection.

Prior Medication:

Excluded:

* Clarithromycin, azithromycin, or ethambutol for more than 10 consecutive days within the 8 weeks prior to study entry OR between the time an initial AFB positive blood sample was collected and study entry.
* Cytokines (other than erythropoietin and interferon-alpha) within 8 weeks prior to study entry.
* Steroids within 8 weeks prior to study entry.
* Cytotoxic chemotherapy within 8 weeks prior to study entry.
* Acute therapy for an AIDS-related opportunistic infection or malignancy, or other acute medical illness or infection within 4 weeks prior to study entry.
* Rifabutin monotherapy if initiated for MAC prophylaxis between the time an initial AFB positive blood sample was collected and study entry.
* Aminoglycosides, quinolones, clofazimine, or rifamycins IF ADMINISTERED IN ANY COMBINATION within 7 days prior to study entry OR between the time an initial AFB positive blood sample was collected and study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hafner R, Study Chair; Drusano G, Study Chair
Locations (8):
- United States (8):
  - Univ of Arizona / Health Science Ctr, Tucson, Arizona
  - Univ of Maryland at Baltimore, Baltimore, Maryland
  - UMDNJ - New Jersey Med School / Cooper Hosp, Camden, New Jersey
  - Albany Med College / Division of HIV Medicine A158, Albany, New York
  - SUNY / Health Sciences Ctr at Stony Brook, Stony Brook, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Richmond AIDS Consortium, Richmond, Virginia